CLINICAL TRIAL: NCT00707278
Title: A Prospective Phase I Study of Radiation Therapy and Concurrent Capecitabine and Oxaliplatin Chemotherapy in the Treatment of Locally Advanced Pancreas Adenocarcinoma
Brief Title: Radiation Therapy and Capecitabine/Oxaliplatin Chemotherapy in the Treatment of Locally Advanced Pancreas Adenocarcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI13633
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Cancer; Pancreas
MeSH Terms: conditions — Neoplasms | interventions — Radiotherapy; Capecitabine; Drug Therapy; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Experimental): All participants enrolled.
  Interventions: Radiation: Radiation Therapy; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Radiation: Radiation Therapy — Radiation therapy will be delivered concurrently with capecitabine and oxaliplatin chemotherapy Radiation therapy dose will be 50.4 Gy (1.8 Gy per day, 5 days per week, for 28 treatments).
Drug: Capecitabine — Capecitabine Dose (given twice daily concurrent with radiation therapy) Dose level 1: 400 mg/m2 Dose level 2:600 mg/m2 Dose level 3:600 mg/m2
  Other Names: Chemotherapy
Drug: Oxaliplatin — Oxaliplatin Dose (given weekly concurrent with radiation therapy) Dose level 1: 50 mg/m2 Dose level 2: 50 mg/m2 Dose level 3: 60 mg/m2
  Other Names: chemotherapy

SUMMARY:
The study is a prospective phase I trial of radiation therapy concurrent with capecitabine and oxaliplatin chemotherapy in the treatment of locally advanced pancreas adenocarcinoma. Eligibility criteria include pathologically confirmed, non-metastatic adenocarcinoma of the pancreas that is surgically unresectable. Patients will undergo radiation therapy (28 treatments of 1.8 Gy for a total of 50.4 Gy) concurrent with capecitabine and oxaliplatin chemotherapy. The primary objective of the study is to determine the maximum tolerated doses of capecitabine and oxaliplatin when delivered concurrently with 50.4 Gy radiation therapy with or without surgery in this patient population.

Secondary objectives of the study are to determine the tumor response rate, survival rate, local control rate and the rate of distant metastases following capecitabine, oxaliplatin, and radiation therapy with or without surgery and to determine the rate at which patients with unresectable disease become resectable.

DETAILED DESCRIPTION:
Patients will undergo radiation therapy (28 treatments of 1.8 Gy for a total of 50.4 Gy) concurrent with capecitabine and oxaliplatin chemotherapy. The primary objective of the study is to determine the maximum tolerated doses of capecitabine and oxaliplatin when delivered concurrently with 50.4 Gy radiation therapy with or without surgery in this patient population.

Three dose levels are planned, as shown in the "Dose Escalation" table below. Three patients are planned at each level. When 3 patients have completed an entire chemoradiation course and are monitored for at least 2 weeks after the end of treatment without the occurrence of dose limiting toxicities (DLTs), then the next 3 patients will be treated at the next highest dose level. If one of the first three patients treated at any given dose level experiences a DLT, three further patients will be treated at that level. If only one in six patients at a given level experiences a DLT, escalation can proceed. If two or more of three to six patients at the lowest administered dose level experience DLTs, then the MTD is below the lowest administered dose, but no specific MTD will be defined. If two or more of three to six patients at a higher dose level experiences DLTs, the dose preceding the lowest dose level satisfying this criterion will be declared the MTD. If all the dose levels are exhausted without two or more of three to six patients experiencing DLTs, then the MTD is higher than the maximum administered dose, but no specific MTD will be defined. If MTD is reached at a given dose level, then additional patients can be accrued to the next lowest dose level, such that up to six patients can be accrued to the dose level below MTD. Because three dose levels are planned, with 3 to 6 patients enrolled in each dose level, a minimum of 9 and a maximum of 18 patients are required for trial completion.

ELIGIBILITY:
Patient Selection Criteria

* Pathologically confirmed adenocarcinoma of the pancreas.
* No distant metastases (no metastases beyond regional lymph nodes).
* Deemed surgically unresectable by a surgical oncologist due to hepatic artery, celiac axis, superior mesenteric artery, superior mesenteric vein, portal vein, aorta, inferior vena cava, and/or rib/vertebral body involvement as defined by CT/MRI scan and/or endoscopic ultrasound (EUS).
* No malignancy (within the past two years) except for non-melanomatous skin cancer or carcinoma in situ of the cervix, uterus, or bladder.
* No previous chemotherapy for pancreatic cancer.
* No prior irradiation to the planned field.
* Zubrod performance status 0-1.
* Granulocytes > 1,800, platelets > 100,000/ul, bilirubin < 2.0 mg/dL, ALT < 3x upper limits of normal, creatinine < 3.0 mg/dL.
* No significant infection or other coexistent medical condition.
* No pregnant or lactating women.
* Age > 18 years old.
* Signed study-specific consent form prior to registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated doses of capecitabine and oxaliplatin when delivered concurrently with 50.4 Gy radiation therapy with or without surgery in patients with locally advanced pancreas adenocarcinoma. | September 2012

SECONDARY OUTCOMES:
To determine tumor response rate, survival rate, local control rate and rate of distant metastases following capecitabine, oxaliplatin, and radiation therapy with or without surgery in patients with locally advanced pancreas adenocarcinoma. | September 2012

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Shrieve, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States